CLINICAL TRIAL: NCT01722266
Title: Liraglutide in the Treatment of Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University at Buffalo (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Paresh Dandona, Distinguished Professor of Medicine, University at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NN1962
Record Dates: First submitted 2012-11-02; First posted 2012-11-06 (Estimated); Results first posted 2015-03-13 (Estimated); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Type 1 Diabetes
Keywords: Liraglutide; Glucagon; Systolic blood pressure; Weight; Carbohydrate intake; Insulin dose; HbA1c; Post-prandial glucagon
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Body Weight | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Daily Injection
  Interventions: Drug: Placebo
- Liraglutide 1.8mg (Active Comparator): Daily Injection
  Interventions: Drug: Liraglutide
- Liraglutide 1.2mg (Active Comparator): Daily injections
  Interventions: Drug: Liraglutide
- Liraglutide 0.6 mg (Active Comparator): Daily injection
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Liraglutide — Patients randomized to 1.2 mg of liraglutide : They will start liraglutide 0.6 mg sc once daily for one week and will increase the dose to 1.2 mg sc once daily thereafter.
  Patients randomized to 1.8 mg of liraglutide: They will start liraglutide 0.6 mg sc once daily for one week; will increase to 1.2 mg sc once daily for second week and will stay on 1.8 mg of liraglutide from third week onwards.
  Other Names: Victoza
  Arms: Liraglutide 0.6 mg; Liraglutide 1.2mg; Liraglutide 1.8mg
Drug: Placebo — Patients randomized to 1.2 mg of placebo: They will start placebo 0.6 mg sc once daily for one week and then increase to 1.2 mg once daily thereafter.
  Patients randomized to 1.8 mg of placebo: They will start placebo 0.6 mg sc once daily for one week; increase to 1.2 mg sc once daily for second week and then to 1.8 mg sc once daily from third week onwards.
  Arms: Placebo

SUMMARY:
Hypothesis 1: Treatment with Liraglutide in patients with type 1 diabetes decreases fasting, postprandial and the overall mean glucose concentrations.

Aim 1.1: To compare the mean fasting, the mean weekly glucose and the standard deviation of weekly blood glucose concentrations as recorded by continuous glucose monitoring prior to and following 6 weeks and 12 weeks of treatment with 0.6, 1.2 and 1.8 mg of liraglutide daily. In addition, the time spent at glucose concentrations >150 and 200mg/dl and <70 and <40 mg/dl will also be compared.

Aim 1.2: To compare the postprandial glucose concentrations following a test meal before and after 12 weeks of treatment with 0.6, 1.2 and 1.8 mg of liraglutide daily. Glucose concentrations will be measured as areas under the curve for the data obtained from the meal challenge.

Aim 1.3: To compare HbA1c levels(glycated hemoglobin) before and after 12 weeks of treatment with 0.6, 1.2 and 1.8 mg of liraglutide daily Hypothesis 2: Treatment with Liraglutide in patients with type 1 diabetes decreases postprandial glucagon concentrations and increases postprandial C-peptide concentrations.

Aim 2.1: To compare fasting and postprandial glucagon and C-peptide concentrations following a test meal before and after 12 weeks of treatment with 0.6, 1.2 and 1.8 mg of liraglutide daily.

Hypothesis 3: Treatment with Liraglutide in patients with type 1 diabetes delays gastric emptying.

Aim 3.1: To compare the gastric emptying as measured by acetaminophen absorption before and after 12 weeks of treatment with 0.6, 1.2 and 1.8 mg of liraglutide daily.

DETAILED DESCRIPTION:
RESEARCH DESIGN AND METHODS This investigation will be a prospective, randomized, double blind, placebo controlled study conducted in type 1 diabetics. The study will be conducted at Diabetes - Endocrinology Center of WNY at Millard Fillmore Hospital, affiliated to the State University of New York at Buffalo.

Study Population: Seventy two patients with type 1 diabetes on treatment with either continuous subcutaneous insulin infusion (CSII; also known as insulin pump) or multiple (four or more) injections of insulin per day will be included in the study. They will be randomized into 4 groups of 18 patients each. The patients will be randomized to placebo or 0.6 mg, 1.2 mg or 1.8 mg liraglutide daily. In view of the possibility of hypoglycemia and the side effect of nausea all patients will be started on 0.6 mg of liraglutide per day. The dose will then be titrated up to 1.2 and 1.8 mg on a weekly basis. No increases will be made once the target dose has been achieved in each group. Subjects will be recruited from our own patients, our existing database and from advertisements. The following insulin preparations will be used in the study: insulin detemir, glargine, aspart, glulisine and lispro. Subjects will continue to obtain their insulin supplies from their respective pharmacies.

STUDY DESIGN:

Screening Day (day -14):- Each patient will have completed the following procedures prior to participating in the study.

1. Medical History;
2. Physical Exam;
3. Informed consent.
4. Baseline lab draw to measure Complete blood count, comprehensive metabolic panel, Hba1c and lipid profile. All labs will be drawn in the fasting state in the morning before 10am.

Randomization Visit (day -7)

Randomization Method: After the screening visit, subjects who meet the inclusion and exclusion criteria, will be assigned a number by a computerized random number generation program (Microsoft office - Excel) and randomized to receive subcutaneous injection daily of either Liraglutide 0.6mg (18 subjects), 1.2 mg (18 subjects), 1.8 mg (18 subjects) or placebo (18 subjects) for 12 weeks. The subjects and the study coordinators will be blinded to the treatment. The Liraglutide/placebo will be administered via a pen kit (obtained from Novo Nordisk Pharmaceuticals). The dose will be given in the morning. The sponsor is providing study medication in blinded form.

All subjects will be instructed by the study staff in the dosing and administration of the study medication and will be seen by a Certified Diabetes Educator for instruction on injection technique. All subjects will also be seen by a registered dietitian who will review their carbohydrate counting and diet and make an assessment of their calorie and carbohydrate intake. The subjects will be randomized but will not start the placebo or liraglutide injection till study intervention visit 1.

All subjects will be advised to monitor their capillary blood glucose by fingerstick before and 2 hours after each meal and to wear their CGM constantly for the duration of the study The subjects will be asked to keep a diary of their food intake to measure their calorie intake. For the entire duration of the study, the patients will maintain a diary to record any hypoglycemia and other untoward side effects like nausea, changes in appetite and other experiences. Patients will be instructed to call the Diabetes Center or an endocrinology fellow directly in case of any problem or untoward side effects. They will be specifically asked to call if they have hypoglycemia (blood sugar <70 mg/dl) or hyperglycemia (blood sugar >250 mg/dl) on more than one occasion.

Study Intervention Visit 1 day 0:- Subjects will come fasting for this visit. Records of blood glucose concentrations monitored by fingerstick and CGM for the previous 7 days will be obtained to assess their glycemic control prior to liraglutide treatment. They will undergo a meal challenge test (described below), Liraglutide or placebo injections at a dose of 0.6 mg per day will then be started. No reduction will be made in the dose of pre-prandial insulin boluses and basal insulin if A1C is greater than or equal to 7.5%. Subjects will decrease the dose of pre-prandial insulin boluses by 25% and the basal by 25% if their A1C is less than or equal to 7%. Subjects will decrease the dose of pre-prandial insulin boluses and basal insulin by 10% if the A1C is between 7 and & 7.5%. This reduction is based on our experience (see preliminary data). Careful adjustments will be made to insulin doses at the discretion of the investigators on the basis of the glucose data obtained from the patients. The target blood glucose will be preprandial 90-120mg/dl and 2hour PP < 140mg/dl, without increasing the incidence of blood glucose < 70mg/dl. Patients will return to the center after 7 days

Study Intervention Visit 2 day 7:- Blood glucose concentrations will be reviewed. Insulin dose will be adjusted at the discretion of the study investigator to optimize blood sugar control as per the targets mentioned above on day 0 visit. Patients will be advised to increase the Liraglutide dose to 1.2 mg a day in those whose target dose is 1.2 or 1.8 mg. They will return in 7 days.

Study Intervention Visit 3 day 14:- Blood glucose concentrations will be reviewed. Insulin dose will be adjusted at the discretion of the study investigator to optimize blood sugar control as per the targets mentioned above on day 0 visit. Patients with a target dose of 1.8 mg will be advised to increase the dose while others will continue on their previous dose. They will return in 7 days.

Study Intervention Visit 4 day 21, Visit 5 day 28:

Records of blood glucose concentrations of the last 7 days will be collected. Insulin dose will be adjusted at the discretion of the study investigator to optimize blood sugar control as per the targets mentioned above on day 0 visit.

Study Intervention Visit 6 day 42, Visit 7 day 56, Visit 8 day 70:

Records of blood glucose concentrations of the last 15 days will be collected. Insulin dose will be adjusted at the discretion of the study investigator to optimize blood sugar control as per the targets mentioned above on day 0 visit.

Study Intervention Visit 9 day 84 Subjects will come fasting for this visit. Records of blood glucose concentrations monitored by fingerstick or CGM for the previous 7 days will be obtained to assess their glycemic control. They will undergo meal challenge test (described below). After this visit, subjects will be discharged from the study.

Meal challenge test:- In order to assess the changes induced by liraglutide, a meal challenge will be carried out prior to and following liraglutide (day 0 and day 84). (910 Calorie High fat High carbohydrate meal as in several of our previous papers). Acetaminophen (1000 mg for body weight <70 kg or 1500 mg for body weight >70 kg) will be ingested at the beginning of the meal, and the blood levels of acetaminophen will be determined at intervals for assessment of the rate of gastric emptying. Bolus Insulin will be injected immediately before the meal based on the insulin carbohydrate ratio and correction factor for each individual subject. Liraglutide will be injected only on day 84 (45 min prior to the meal). Sequential blood samples will be obtained at 0, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240 and 300 min. Samples at 15, 30, 45, 90, 150 and 210 min will be 5 ml while those at 0, 60, 120, 180, 240 and 300 min will be 30 ml (total volume=210 ml). Blood will be collected from an indwelling intravenous canula in a superficial forearm vein.

Data safety and monitoring:

Timely, accurate, and complete reporting and analysis of safety information obtained from clinical trials are crucial for the protection of subjects and investigators.

All subjects will be referred to liraglutide's labeling safety information, and will be provided a copy of the package insert of the medication. Discussion of the potential side effects and the different warning and precautions will take place at the time of signing the informed consent.

The following Information from the boxed warning in the package insert regarding the risk of thyroid c-cell tumors will be discussed in details with all participating subjects "Liraglutide causes dose-dependent and treatment-duration-dependent thyroid C-cell tumors at clinically relevant exposures in both genders of rats and mice. It is unknown whether Liraglutide causes thyroid C-cell tumors, including medullary thyroid carcinoma (MTC), in humans, as human relevance could not be ruled out by clinical or nonclinical studies. Liraglutide is contraindicated in patients with a personal or family history of MTC and in patients with Multiple Endocrine Neoplasia syndrome type 2 (MEN 2). Based on the findings in rodents, monitoring with serum calcitonin or thyroid ultrasound was performed during clinical trials, but this may have increased the number of unnecessary thyroid surgeries. It is unknown whether monitoring with serum calcitonin or thyroid ultrasound will mitigate human risk of thyroid C-cell tumors."

In addition, the following FDA text regarding the risk of developing fibrosarcomas will be discussed with all participating subjects "In a 2-year repeat subcutaneous dose carcinogenicity study of liraglutide injected once a day in CD-1 mice, a treatment-related increase in fibrosarcomas was seen on the dorsal skin and subcutis, the body surface used for drug injection, in males in the 3 mg/kg/day group. These fibrosarcomas were attributed to the high local concentration of drug near the injection site. The liraglutide concentration in the clinical formulation (6 mg/mL) is 10 times higher than the concentration in the formulation used to administer 3 mg/kg/day liraglutide to mice in the carcinogenicity study (0.6 mg/mL)".

All Adverse events(AEs) will be reported at the time of the visit or by telephone when it occurs. Those meeting the definition of Serious Adverse Events(SAE's) must be reported using the SAE Form. Medical events that occur between the signing of the Informed Consent and the first intake of study drug will be documented in the medical history. Subjects should voluntarily report any AEs or in response to general, non-directed questioning. For each AE volunteered by the subject, the investigator will obtain all the information required to complete the AE page of the Case Report Form(CRF), in accordance with the guidelines that accompany it.

All AEs, regardless of seriousness, severity, or presumed relationship to study therapy, will be recorded using medical terminology in the source document and on the CRF. Whenever possible, diagnoses will be given when signs and symptoms are due to a common etiology (e.g., cough, runny nose, sneezing, sore throat, and head congestion should be reported as "upper respiratory infection). Investigators will record on the CRF their opinion concerning the relationship of the AE to study therapy. All measures required for AE management will be recorded in the source document and reported according to sponsor instructions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with type 1 diabetes mellitus: Fasting c-peptide < 0.1nmol/l on insulin therapy for more than 12 months with or without history of diabetic ketoacidosis.
2. Using a continuous glucose monitoring device (CGM) and regularly measuring their blood sugars four times daily
3. HbA1c of less than 8.5%.
4. Well versed with carbohydrate counting
5. Age 18-75 years

Exclusion Criteria:

1. Type 1 diabetes for less than 12 months;
2. Coronary event or procedure (myocardial infarction, unstable angina, coronary artery bypass, surgery or coronary angioplasty) in the previous four weeks;
3. Hepatic disease (transaminase > 3 times normal) or cirrhosis;
4. Renal impairment (serum creatinine > 1.5);
5. HIV or Hepatitis C positive status;
6. Participation in any other concurrent clinical trial;
7. Any other life-threatening, non-cardiac disease;
8. Use of an investigational agent or therapeutic regimen within 30 days of study.
9. history of pancreatitis
10. pregnancy
11. inability to give informed consent
12. history of gastroparesis
13. history of medullary thyroid carcinoma or MEN 2 syndrome.
14. Family history of MEN 2, Family history of medullary thyroid cancer, or familial medullary thyroid cancer
15. Women of childbearing potential who are not using adequate contraception 16) Women who are pregnant

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-11-01 (Actual); Primary Completion 2014-04-01 (Actual); Study Completion 2014-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paresh Dandona, MBBS, PhD, Principal Investigator — Kaleida Health
Locations (1):
- Diabetes-Endocrinology Center of Western NY, Williamsville, New York, United States

REFERENCES:
- [Background] Kuhadiya ND, Malik R, Bellini NJ, Patterson JL, Traina A, Makdissi A, Dandona P. Liraglutide as additional treatment to insulin in obese patients with type 1 diabetes mellitus. Endocr Pract. 2013 Nov-Dec;19(6):963-7. doi: 10.4158/EP13065.OR. PMID 23807520
- [Background] Varanasi A, Bellini N, Rawal D, Vora M, Makdissi A, Dhindsa S, Chaudhuri A, Dandona P. Liraglutide as additional treatment for type 1 diabetes. Eur J Endocrinol. 2011 Jul;165(1):77-84. doi: 10.1530/EJE-11-0330. Epub 2011 Jun 6. PMID 21646283
- [Background] Kielgast U, Asmar M, Madsbad S, Holst JJ. Effect of glucagon-like peptide-1 on alpha- and beta-cell function in C-peptide-negative type 1 diabetic patients. J Clin Endocrinol Metab. 2010 May;95(5):2492-6. doi: 10.1210/jc.2009-2440. Epub 2010 Mar 5. PMID 20207828
- [Background] Rother KI, Spain LM, Wesley RA, Digon BJ 3rd, Baron A, Chen K, Nelson P, Dosch HM, Palmer JP, Brooks-Worrell B, Ring M, Harlan DM. Effects of exenatide alone and in combination with daclizumab on beta-cell function in long-standing type 1 diabetes. Diabetes Care. 2009 Dec;32(12):2251-7. doi: 10.2337/dc09-0773. Epub 2009 Oct 6. PMID 19808924
- [Background] Ghanim H, Aljada A, Daoud N, Deopurkar R, Chaudhuri A, Dandona P. Role of inflammatory mediators in the suppression of insulin receptor phosphorylation in circulating mononuclear cells of obese subjects. Diabetologia. 2007 Feb;50(2):278-85. doi: 10.1007/s00125-006-0508-9. Epub 2006 Dec 16. PMID 17180352
- [Background] Wajchenberg BL, Feitosa AC, Rassi N, Lerario AC, Betti RT. Glycemia and cardiovascular disease in type 1 diabetes mellitus. Endocr Pract. 2008 Oct;14(7):912-23. doi: 10.4158/EP.14.7.912. PMID 18996824
- [Background] Buse JB, Klonoff DC, Nielsen LL, Guan X, Bowlus CL, Holcombe JH, Maggs DG, Wintle ME. Metabolic effects of two years of exenatide treatment on diabetes, obesity, and hepatic biomarkers in patients with type 2 diabetes: an interim analysis of data from the open-label, uncontrolled extension of three double-blind, placebo-controlled trials. Clin Ther. 2007 Jan;29(1):139-53. doi: 10.1016/j.clinthera.2007.01.015. PMID 17379054
- [Background] Montanya E, Sesti G. A review of efficacy and safety data regarding the use of liraglutide, a once-daily human glucagon-like peptide 1 analogue, in the treatment of type 2 diabetes mellitus. Clin Ther. 2009 Nov;31(11):2472-88. doi: 10.1016/j.clinthera.2009.11.034. PMID 20109994
- [Background] Varanasi A, Patel P, Makdissi A, Dhindsa S, Chaudhuri A, Dandona P. Clinical use of liraglutide in type 2 diabetes and its effects on cardiovascular risk factors. Endocr Pract. 2012 Mar-Apr;18(2):140-5. doi: 10.4158/EP11169.OR. PMID 21856595
- [Background] Varanasi A, Chaudhuri A, Dhindsa S, Arora A, Lohano T, Vora MR, Dandona P. Durability of effects of exenatide treatment on glycemic control, body weight, systolic blood pressure, C-reactive protein, and triglyceride concentrations. Endocr Pract. 2011 Mar-Apr;17(2):192-200. doi: 10.4158/EP10199.OR. PMID 20841306
- [Background] Okerson T, Yan P, Stonehouse A, Brodows R. Effects of exenatide on systolic blood pressure in subjects with type 2 diabetes. Am J Hypertens. 2010 Mar;23(3):334-9. doi: 10.1038/ajh.2009.245. Epub 2009 Dec 17. PMID 20019672
- [Background] Lebovitz HE. Adjunct therapy for type 1 diabetes mellitus. Nat Rev Endocrinol. 2010 Jun;6(6):326-34. doi: 10.1038/nrendo.2010.49. Epub 2010 Apr 20. PMID 20404854
- [Derived] Kuhadiya ND, Dhindsa S, Ghanim H, Mehta A, Makdissi A, Batra M, Sandhu S, Hejna J, Green K, Bellini N, Yang M, Chaudhuri A, Dandona P. Addition of Liraglutide to Insulin in Patients With Type 1 Diabetes: A Randomized Placebo-Controlled Clinical Trial of 12 Weeks. Diabetes Care. 2016 Jun;39(6):1027-35. doi: 10.2337/dc15-1136. Epub 2016 Apr 5. PMID 27208343

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Daily Injection
  Placebo: Patients randomized to 1.2 mg of placebo: They will start placebo 0.6 mg sc once daily for one week and then increase to 1.2 mg once daily thereafter.
  Patients randomized to 1.8 mg of placebo: They will start placebo 0.6 mg sc once daily for one week; increase to 1.2 mg sc once daily for second week and then to 1.8 mg sc once daily from third week onwards.
- Liraglutide 1.8mg; Liraglutide 0.6 mg: Daily Injection
  Liraglutide: Patients randomized to 1.2 mg of liraglutide : They will start liraglutide 0.6 mg sc once daily for one week and will increase the dose to 1.2 mg sc once daily thereafter.
  Patients randomized to 1.8 mg of liraglutide: They will start liraglutide 0.6 mg sc once daily for one week; will increase to 1.2 mg sc once daily for second week and will stay on 1.8 mg of liraglutide from third week onwards.
- Liraglutide 1.2mg: Daily injections
  Liraglutide: Patients randomized to 1.2 mg of liraglutide : They will start liraglutide 0.6 mg sc once daily for one week and will increase the dose to 1.2 mg sc once daily thereafter.
  Patients randomized to 1.8 mg of liraglutide: They will start liraglutide 0.6 mg sc once daily for one week; will increase to 1.2 mg sc once daily for second week and will stay on 1.8 mg of liraglutide from third week onwards.
Period: Overall Study
Arm/Group | Placebo | Liraglutide 1.8mg | Liraglutide 1.2mg | Liraglutide 0.6 mg
Started | 18 | 18 | 18 | 18 (3 withdrew consent; 1 dropped out due to nausea)
Completed | 17 | 15 | 13 | 18 (3 subjects randomized to 1.2 mg group and 1 to 1.8 mg group tolerated only 0.6 mg)
Not Completed | 1 | 3 | 5 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0
Not completed — Tolerated only 0.6 mg liraglutide | 0 | 1 | 3 | 0
Not completed — Dropped out due to Nausea | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Liraglutide 1.8mg | Liraglutide 1.2mg | Liraglutide 0.6 mg | Total
Number analyzed (Participants) | 17 | 15 | 13 | 18 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (3) | 42 (3) | 42 (3) | 45 (4) | 44 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 5 | 9 | 35
  Male | 7 | 4 | 8 | 9 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 0 | 2
  White | 14 | 15 | 13 | 17 | 59
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 15 | 13 | 18 | 63
Age of Type 1 Diabetes Diagnosis [Mean (Standard Deviation); unit: years] | 19 (3) | 21 (3) | 21 (3) | 19 (3) | 20 (1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Weekly Glucose Concentrations
Description: The primary endpoint of the study is to detect a difference from baseline in mean weekly blood glucose concentrations before and after 12 weeks of treatment in each of the Liraglutide groups.
Time Frame: 12 Weeks
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Placebo | Liraglutide 1.8mg | Liraglutide 1.2mg | Liraglutide 0.6 mg
Number analyzed (Participants) | 17 | 15 | 13 | 18
mg/dl | 1 (0) | -10 (1) | -10 (2) | -0.3 (2)

2. Secondary Outcome: Change in HbA1c
Description: Change from baseline (week 0) in HbA1c at 12 weeks after treatment
Time Frame: 12 Weeks
Measure: Mean (Standard Error); unit: Percent of Hemoglobin (%)
Arm/Group | Placebo | Liraglutide 1.8mg | Liraglutide 1.2mg | Liraglutide 0.6 mg
Number analyzed (Participants) | 17 | 15 | 13 | 18
Percent of Hemoglobin (%) | -0.30 (0.15) | -0.42 (0.15) | -0.78 (0.15) | -0.26 (0.17)

3. Secondary Outcome: Change in Body Weight From Baseline
Description: Change in Body weight in Kg from baseline after 12 weeks of treatment
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: Kg
Arm/Group | Placebo | Liraglutide 1.8mg | Liraglutide 1.2mg | Liraglutide 0.6 mg
Number analyzed (Participants) | 17 | 15 | 13 | 18
Kg | -0.3 (0.5) | -4.8 (0.7) | -5.0 (1.2) | -2.7 (0.6)

4. Secondary Outcome: Change in Total Insulin Dose From Baseline
Description: Total daily insulin dose = Basal insulin dose plus bolus insulin dose. Change from baseline in Total daily insulin dose at 12 weeks from treatment.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: Units of insulin
Arm/Group | Placebo | Liraglutide 1.8mg | Liraglutide 1.2mg | Liraglutide 0.6 mg
Number analyzed (Participants) | 17 | 15 | 13 | 18
Units of insulin | -3.4 (0.7) | -10 (0.5) | -12.1 (0.7) | -2.8 (0.7)

5. Secondary Outcome: Change in the Area Under Curve (AUC) of Glucose Following the Meal
Description: Change in the Area Under Curve (AUC0h-5h) of glucose concentration measured following meal challenge of up to 5hrs performed at baseline (week 0) at 12 weeks following treatment.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: g * 5 h * dL^-1
Arm/Group | Placebo | Liraglutide 1.8mg | Liraglutide 1.2mg | Liraglutide 0.6 mg
Number analyzed (Participants) | 17 | 15 | 13 | 18
g * 5 h * dL^-1 | 0.04 (0) | -0.55 (10) | -0.55 (10) | -0.01 (0.11)

6. Secondary Outcome: Change in Carbohydrate Intake
Description: Change from baseline (0 week) in Daily Carbohydrate intake (in grams) at 12 weeks after treatment.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: grams
Arm/Group | Placebo | Liraglutide 1.8mg | Liraglutide 1.2mg | Liraglutide 0.6 mg
Number analyzed (Participants) | 17 | 15 | 13 | 18
grams | -13.4 (2.6) | -46.4 (1.6) | -47.6 (2.6) | -23.7 (2.5)

7. Secondary Outcome: Change in Glucagon Concentrations
Description: change from baseline (week 0) in glucagon concentrations following 12 weeks of treatment
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: ng/L
Arm/Group | Placebo | Liraglutide 1.8mg | Liraglutide 1.2mg | Liraglutide 0.6 mg
Number analyzed (Participants) | 17 | 15 | 13 | 18
ng/L | 5 (3) | 9 (6) | -6 (9) | 7 (4)

ADVERSE EVENTS:
Time Frame: 12 weeks.
Arm/Group | Placebo | Liraglutide 1.8mg | Liraglutide 1.2mg | Liraglutide 0.6 mg
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/15 | 0/13 | 0/18
Other Adverse Events (participants affected / at risk) | 3/17 | 9/15 | 10/13 | 11/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=17) | Liraglutide 1.8mg (N=15) | Liraglutide 1.2mg (N=13) | Liraglutide 0.6 mg (N=18)
Transient Nausea (Gastrointestinal disorders) | 3 (3) | 9 (9) | 10 (10) | 11 (11) — Transient nausea reported at the time of initiation of liraglutide for first 2-5 days and then another 2-4 days at the time of escalation of the dose. Nausea is a common side effect of liralgutide.

LIMITATIONS AND CAVEATS:
Three subjects randomized to 1.2 mg group and one subject randomized to 1.8 mg group tolerated only 0.6 mg. These 4 subjects were included in the 0.6 mg group for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No